CLINICAL TRIAL: NCT01511562
Title: A Randomized Phase II Trial of Myeloablative Versus Non-Myeloablative Consolidation Chemotherapy for Newly Diagnosed Primary CNS B-cell Lymphoma
Brief Title: Combination Chemotherapy With or Without Autologous Stem Cell Transplant in Treating Patients With Central Nervous System B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-51101; CALGB-51101; CDR0000721927 (Registry Identifier: NCI Physician Data Query); NCI-2012-00110 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2012-01-13; First posted 2012-01-18 (Estimated); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Carmustine; Cytarabine; Etoposide; Thiotepa; Stem Cell Transplantation; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Other): Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo stem cell transplant.
  Interventions: Drug: carmustine; Drug: thiotepa; Procedure: stem cell transplant; Drug: G-CSF
- Arm II (Other): Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo consolidation chemotherapy.
  Interventions: Drug: cytarabine; Drug: etoposide; Drug: G-CSF

INTERVENTIONS:
Drug: carmustine — Given IV
  Arms: Arm I
Drug: cytarabine — Given IV
  Arms: Arm II
Drug: etoposide — Given IV
  Arms: Arm II
Drug: thiotepa — Given IV
  Arms: Arm I
Procedure: stem cell transplant
  Arms: Arm I
Drug: G-CSF

SUMMARY:
The purpose of this study is to find out what effects (good and/or bad) treatment with chemotherapy and stem cell transplant compared with chemotherapy alone will have on primary CNS B-cell lymphoma. Currently the best treatment for patients with primary CNS B-cell lymphoma is not known.

DETAILED DESCRIPTION:
Primary Objective:

To compare the two-year progression-free survival (PFS) of patients treated with the myeloablative consolidation treatment strategy of HDT/ASCT versus those treated with non-myeloablative consolidation chemotherapy with cytarabine and etoposide

Secondary Objectives:

1. To compare the two-year event-free survival (EFS) of patients treated with consolidation HDT/ASCT versus those treated with consolidation chemotherapy consisting of etoposide and cytarabine
2. To compare the overall survival (OS) of patients treated with the consolidation HDT/ASCT versus those treated with consolidation chemotherapy consisting of etoposide and cytarabine
3. To assess the toxicities associated with consolidation HDT/ASCT versus consolidation consisting of etoposide and cytarabine
4. To determine diffusion MRI metrics (ADCmini, ADC25%, and ADCmean) prior to induction chemotherapy, after one full induction chemotherapy cycle, and at the end of induction chemotherapy as a predictor of response and outcome (CALGB 581101)
5. To determine brain FDG-PET metrics (tumor SUV and tumor versus background SUV) prior to induction chemotherapy, after one full induction chemotherapy cycle, and at the end of induction chemotherapy as a predictor of response and outcome (CALGB 581101)
6. To determine whether low baseline ADC measurements are associated with shorter PFS and OS (CALGB 581101)
7. To determine whether reduction in tumor SUV by > 25% on brain FDG-PET/CT after one cycle of induction therapy is associated with improved PFS and OS (CALGB 581101)
8. To determine which IHC-based biomarkers are predictive of an adverse prognosis (CALGB 151113)
9. To determine which IHC-based biomarkers are predictive of a favorable prognosis (CALGB 151113) for BCL6 (B-cell CLL/lymphoma 6), and STAT 6 (signal transducer and activator of transcription 6, interleukin-4 induced)
10. To analyze tumor tissue for gene expression profiles, and to correlate these profiles with treatment outcomes (CALGB 151113)
11. To determine whether CSF proteome is a predictor of outcomes (prognostic marker) irrespective of treatment arm (CALGB 151113) for (IL-10 (interleukin 10) and C3 (complement component 3)
12. To assess the neurocognitive function of patients treated with consolidation HDT/ASCT versus those treated with consolidation chemotherapy (etoposide and cytarabine) as measured by serial administration of the International PCNSL Collaborative Group (IPCG) neurocognitive battery and evaluate the long-term survivorship differences between the two arms (CALGB 71105)

ELIGIBILITY:
1. Documentation of Disease: Diagnosis of primary CNS diffuse large B-cell lymphoma confirmed by one of the following: brain biopsy or resection, cerebrospinal fluid and vitreous fluid.
2. Other Lymphomas: Patients must have no evidence or history of non-Hodgkin lymphoma (NHL) outside of CNS.
3. Previous Treatment: Patients must have no prior chemotherapy or radiation therapy for lymphoma.
4. Age- Patients must be between the ages of 18 and 75 years.
5. Karnofsky Performance Scale - Patients must measure Karnofsky Performance Scale ≥ 30 (≥ 50 for patients ages 60-70).
6. Pregnancy and Nursing Status - Patients must be non-pregnant and non-nursing; women of childbearing potential must have a negative serum or urine pregnancy test 10-14 days prior to registration; in addition, women and men of childbearing potential must commit to use an effective form of contraception throughout their participation in this study; appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom)
7. HIV - Patients must have negative HIV serology.
8. Hepatitis - Patients must have negative HCV serology (unless HBsAb positive patient has recently received HBV vaccine, in this case HBcAb should be negative). All patients must be screened for hepatitis B infection before starting treatment. Those patients who test positive for hepatitis B should be closely monitored for evidence of active HBV infection and hepatitis during and for several months after rituximab treatment. PCNSL patients with a history of hepatitis B infection should be treated with entecavir or lamivudine (physician discretion for choice of drug) as antiviral prophylaxis to prevent hepatitis B reactivation.
9. Organ Transplant or Immunosuppressant Therapy - Patient must have no history of organ transplantation or ongoing immunosuppressant therapy.
10. Required Initial Laboratory Values: ANC ≥ 1500/mcL, AST and ALT < 2 x upper limit of normal (ULN), total bilirubin ≤ 3 mg/dL, creatinine clearance ≥ 50 mL/min, platelet count ≥ 100,000/mcL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-09; Primary Completion 2020-12-10 (Actual); Study Completion 2027-05-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, MPH, Study Chair — Massachusetts General Hospital
Locations (126):
- United States (126):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Reid Health, Richmond, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Surgical Associates Inc, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Batchelor TT, Giri S, Ruppert AS, Geyer SM, Smith SE, Mohile N, Swinnen LJ, Friedberg JW, Kahl BS, Bartlett NL, Hsi ED, Cheson BD, Wagner-Johnston N, Nayak L, Leonard JP, Rubenstein JL. Myeloablative vs nonmyeloablative consolidation for primary central nervous system lymphoma: results of Alliance 51101. Blood Adv. 2024 Jun 25;8(12):3189-3199. doi: 10.1182/bloodadvances.2023011657. PMID 38598710

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo stem cell transplant.> > carmustine: Given IV>
  > thiotepa: Given IV>
  > stem cell transplant>
  > G-CSF
- Arm II: Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo consolidation chemotherapy.>
  > cytarabine: Given IV>
  > etoposide: Given IV>
  > G-CSF
Period: Induction
Arm/Group | Arm I | Arm II
Started (Eligible and began treatment) | 54 | 54
Completed | 45 | 40
Not Completed | 9 | 14
Not completed — Adverse Event | 2 | 0
Not completed — Disease Progression | 3 | 7
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Other | 3 | 0
Period: Consolidation
Arm/Group | Arm I | Arm II
Started | 38 | 34
Completed | 36 | 34
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Median (Standard Deviation); unit: years] | 58.3 (10.41) | 59.5 (10.76) | 58.9 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 32 | 29 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 47 | 48 | 95
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 49 | 50 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 54 | 54 | 108
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — A standard way of measuring the ability of cancer patients to perform ordinary tasks. The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities.
  Participants
    30 | 1 | 1 | 2
    40 | 0 | 2 | 2
    50 | 4 | 5 | 9
    60 | 6 | 6 | 12
    70 | 12 | 15 | 27
    80 | 13 | 9 | 22
    90 | 17 | 14 | 31
    100 | 1 | 2 | 3
Age and KPS Category [Count of Participants; unit: Participants]
  Age < 51 years and any KPS status | 10 | 10 | 20
  Age >= 51 years and KPS < 70 | 11 | 12 | 23
  Age >= 51 years and KPS >=70 | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The primary endpoint is to compare the two-year progression-free survival (PFS) of patients treated with the myeloablative consolidation treatment strategy of HDT/ASCT versus those treated with non-myeloablative consolidation chemotherapy with cytarabine and etoposide.
  PFS time = time from Registration to earliest date of Progression or Death due to any cause, censoring non-progressed and alive patients at the date of last disease status evaluation.
  Response will be defined using the modified IPCG criteria. Progressive disease is defined as > 25% increase in contrast-enhancing CNS (brain and spine if latter abnormal at baseline) disease, appearance of any new, measurable (>/= 10mm) contrast-enhancing disease or recurrent or new ocular or CSF disease.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants w/out event
Groups:
- Arm I: Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo stem cell transplant.
  >
  > carmustine: Given IV
  >
  > thiotepa: Given IV
  >
  > stem cell transplant
  >
  > G-CSF
- Arm II: Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo consolidation chemotherapy.
  >
  > cytarabine: Given IV
  >
  > etoposide: Given IV
  >
  > G-CSF
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 54 | 54
percentage of participants w/out event | 72.9 [58.5 to 83.0] | 50.6 [36.1 to 63.3]

2. Secondary Outcome: Event Free Survival
Description: To compare the two-year event-free survival (EFS) of patients treated with consolidation HDT/ASCT versus those treated with consolidation chemotherapy consisting of etoposide and cytarabine.
  EFS event = same definition as PFS with non-protocol treatment also considered an event
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants w/out event
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 54 | 54
percentage of participants w/out event | 65.7 [51.2 to 76.9] | 48.5 [34.2 to 61.4]

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Number of patients reporting at least one adverse event at least possibly related to treatment.
Time Frame: 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 54 | 54
Participants | 54 | 53

4. Secondary Outcome: Overall Survival
Description: To compare the overall survival (OS) of patients treated with the consolidation HDT/ASCT versus those treated with consolidation chemotherapy consisting of etoposide and cytarabine.
  OS event = Registration/Randomization to Death due to any cause
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants alive
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 54 | 54
percentage of participants alive | 86.6 [73.9 to 93.4] | 78.3 [64.3 to 87.4]

ADVERSE EVENTS:
Time Frame: 7 years
Groups:
- Arm I: Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo stem cell transplant. > > carmustine: Given IV >
  * thiotepa: Given IV >
  * stem cell transplant >
  * G-CSF
- Arm II: Patients undergo induction therapy for five cycles as defined in the protocol. Patients undergo consolidation chemotherapy. >
  * cytarabine: Given IV >
  * etoposide: Given IV >
  * G-CSF
Arm/Group | Arm I | Arm II
All-Cause Mortality (participants affected / at risk) | 11/54 | 15/54
Serious Adverse Events (participants affected / at risk) | 21/54 | 33/54
Other Adverse Events (participants affected / at risk) | 54/54 | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=54) | Arm II (N=54)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (5)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders and administration site conditions) | 1 (1) | 0 (0)
Sudden death NOS (General disorders and administration site conditions) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 3 (3)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (6)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 4 (7)
Creatinine increased (Investigations) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 5 (6)
Neutrophil count decreased (Investigations) | 5 (5) | 4 (4)
Platelet count decreased (Investigations) | 2 (2) | 4 (4)
White blood cell decreased (Investigations) | 2 (2) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 3 (3)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=54) | Arm II (N=54)
Anemia (Blood and lymphatic system disorders) | 53 (381) | 48 (233)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 9 (13) | 1 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 22 (26) | 15 (17)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (5) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 5 (14) | 7 (10)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 3 (4) | 1 (9)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (2)
Blurred vision (Eye disorders) | 6 (12) | 5 (7)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 2 (3) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (3) | 2 (3)
Flashing lights (Eye disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Night blindness (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2) | 2 (3)
Colitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 17 (33) | 20 (50)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 28 (49) | 18 (29)
Dry mouth (Gastrointestinal disorders) | 2 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 9 (11) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (4) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (3) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 31 (47) | 16 (28)
Nausea (Gastrointestinal disorders) | 34 (97) | 20 (53)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (42) | 17 (25)
Chills (General disorders and administration site conditions) | 7 (7) | 3 (5)
Death NOS (General disorders and administration site conditions) | 0 (0) | 1 (1)
Edema face (General disorders and administration site conditions) | 0 (0) | 2 (2)
Edema limbs (General disorders and administration site conditions) | 13 (29) | 13 (27)
Fatigue (General disorders and administration site conditions) | 38 (125) | 27 (94)
Fever (General disorders and administration site conditions) | 6 (7) | 6 (7)
Gait disturbance (General disorders and administration site conditions) | 22 (77) | 21 (60)
Gen disord and admin site conds-Oth spec (General disorders and administration site conditions) | 2 (7) | 1 (1)
Infusion site extravasation (General disorders and administration site conditions) | 0 (0) | 1 (1)
Injection site reaction (General disorders and administration site conditions) | 1 (1) | 0 (0)
Localized edema (General disorders and administration site conditions) | 1 (3) | 3 (7)
Malaise (General disorders and administration site conditions) | 2 (2) | 1 (1)
Neck edema (General disorders and administration site conditions) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders and administration site conditions) | 3 (3) | 1 (1)
Pain (General disorders and administration site conditions) | 2 (3) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (3) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 7 (7) | 3 (3)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 2 (2)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 3 (4) | 3 (6)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3) | 5 (7)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (9) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (8) | 5 (5)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial throm time prolonged (Investigations) | 2 (2) | 2 (4)
Alanine aminotransferase increased (Investigations) | 47 (171) | 47 (177)
Alkaline phosphatase increased (Investigations) | 13 (27) | 8 (13)
Aspartate aminotransferase increased (Investigations) | 46 (153) | 47 (167)
Blood bilirubin increased (Investigations) | 29 (75) | 28 (61)
CD4 lymphocytes decreased (Investigations) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 35 (125) | 24 (55)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 4 (10) | 1 (1)
Lymphocyte count decreased (Investigations) | 31 (161) | 23 (104)
Lymphocyte count increased (Investigations) | 5 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 46 (144) | 41 (113)
Platelet count decreased (Investigations) | 48 (258) | 49 (182)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (7) | 1 (1)
Weight loss (Investigations) | 8 (15) | 2 (4)
White blood cell decreased (Investigations) | 28 (99) | 23 (65)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 25 (56) | 16 (28)
Dehydration (Metabolism and nutrition disorders) | 5 (8) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2) | 3 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (64) | 22 (71)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5) | 5 (5)
Hypernatremia (Metabolism and nutrition disorders) | 5 (12) | 5 (8)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 27 (72) | 19 (46)
Hypocalcemia (Metabolism and nutrition disorders) | 24 (66) | 18 (50)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 28 (88) | 23 (53)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (17) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 8 (11) | 12 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (22) | 8 (15)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Obesity (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 14 (24) | 6 (9)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (8)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 7 (19) | 7 (12)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 4 (5) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 4 (8) | 6 (7)
Dizziness (Nervous system disorders) | 11 (14) | 4 (5)
Dysarthria (Nervous system disorders) | 5 (13) | 6 (12)
Dysgeusia (Nervous system disorders) | 9 (15) | 2 (4)
Dysphasia (Nervous system disorders) | 2 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 19 (36) | 14 (31)
Hydrocephalus (Nervous system disorders) | 1 (3) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 2 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 9 (15) | 8 (12)
Muscle weakness left-sided (Nervous system disorders) | 1 (4) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 6 (6) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 4 (6) | 2 (5)
Peripheral motor neuropathy (Nervous system disorders) | 2 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (11) | 5 (8)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (5) | 4 (5)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1)
Spasticity (Nervous system disorders) | 1 (3) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 3 (3) | 3 (6)
Anxiety (Psychiatric disorders) | 4 (8) | 4 (8)
Confusion (Psychiatric disorders) | 16 (33) | 18 (40)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2)
Delusions (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (9) | 3 (3)
Hallucinations (Psychiatric disorders) | 1 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 9 (14) | 9 (22)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 8 (15) | 5 (12)
Chronic kidney disease (Renal and urinary disorders) | 2 (7) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (4) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (2) | 2 (7)
Urinary frequency (Renal and urinary disorders) | 2 (5) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (2) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 9 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 7 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (10)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (10) | 5 (7)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 13 (47) | 15 (30)
Hypotension (Vascular disorders) | 8 (9) | 2 (2)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 4 (10) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT01511562/Prot_SAP_000.pdf